CLINICAL TRIAL: NCT04320017
Title: Joint Use of Electrocardiogram and Transthoracic Echocardiography With Other Clinico-biological Parameters in an Observational Study to Monitor Cardio-vascular Events and Predict Outcomes in Patients Diagnosed With COVID-19
Acronym: JOCOVID
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, Head of Investigations in Clinical Investigation Centers Paris-Est, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-20-05
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: COVID-19; Myocardial Injury; Myocarditis
Keywords: Coronavirus; Heart conditions; Cardio-vascular outcomes
MeSH Terms: conditions — COVID-19; Myocarditis; Coronavirus Infections | interventions — Electrocardiography; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 patients: Patients diagnosed with COVID-19 by PCR done on nasal sample.
  Interventions: Diagnostic Test: Electrocardiogram, transthoracic echocardiography and clinico-biological parameters in routine care

INTERVENTIONS:
Diagnostic Test: Electrocardiogram, transthoracic echocardiography and clinico-biological parameters in routine care — * 12 derivations electrocardiogram done at baseline and repeated every 3 days
  * transthoracic echocardiography at baseline
  * clinical features at baseline: WHO performans status comorbidities and treatments
  * biological results in routine care, such as baseline full blood count, inflammation markers: C-reactive protein, procalcitonin, interleukin-6 and ferritin, coagulation and troponin and brain natriuretic peptide

SUMMARY:
COVID-19 outbreak is often lethal. Mortality has been associated with several cardio-vascular risk factors such as diabetes, obesity, hypertension and tobacco use. Other clinico-biological features predictive of mortality or transfer to Intensive Care Unit are also needed. Cases of myocarditis have also been reported with COVID-19.

Cardio-vascular events have possibly been highly underestimated. The study proposes to systematically collect cardio-vascular data to study the incidence of myocarditis and coronaropathy events during COVID-19 infection.We will also assess predictive factors for transfer in Intensive Care Unit or death.

ELIGIBILITY:
Inclusion Criteria:

- COVID-19 positive patients admitted in a ward identified by positive PCR on nasal swab samples

Exclusion Criteria:

- Patients who refused the use of their routine care data after information by investigators.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted in Pitié-Salpêtrière hospital will be eligible, if the electrocardiogram and the transthoracic echocardiography is technically feasible.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Incidence of acute myocardial events in COVID-19 population at baseline and during hospital stay | ECG and concomitant troponine at day 1 after admission at day 1, day 3 day 6 the first week after admission, and then at day 14 and before the patient is discharged (up to 20 days)
  Viral myocarditis or myocardial infarction or stenosis detected with ST segment elevation or depression associated with troponine elevation and transthoracic echocardiography

SECONDARY OUTCOMES:
Description of cardiovascular outcomes in the cohort | During hospital admission (up to 20 days)
  Cardio-vascular events including but not limited to: myocardial infarction or stenosis, stroke, pulmonary embolism, deep vein thrombosis, ventricular dysfunctio, conduction disorders and sudden death
Prognosis role of baseline cardio-vascular caracteristics on patients survival | 1st day of admission
  Biological biomarkers including but not limited to: baseline troponine T, D-dimers, NT-proBNP, creatinine phosphokinase, creatininemia, ionogram, renine-angiotensin aldosterone system profiling, glycemia (fasting), HbA1c, steroid profiling, lipid profiling
Prediction of cardio-vascular events with baseline characteristics | Baseline on first day of admission
Characterization of inflammation on cardio-vascular outcomes | Baseline and at day 3 day 6 day 14 and before patient is discharged (up to 20 days)
  Biological markers including but not limited to: C reactive protein, procalcitonine, fibrinogen, interleukin-6
Prognosis role of baseline clinico-biological caracteristics on patients transfer to ICU and survival | Baseline and at day 3 day 6 day 14 and before patient is discharged (up to 20 days)
  clinical features at baseline: WHO performans status comorbidities and treatments Biological markers including but not limited to: full blood count, C reactive protein, procalcitonine, fibrinogen, interleukin-6, troponin and brain natriuretic peptide

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Investigation Center Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fenioux C, Allenbach Y, Vozy A, Salem JE, Maalouf G, Vieira M, Le Joncour A, Benveniste O, Saadoun D, Frere C, Campedel L, Salem P, Gligorov J, Funck-Brentano C, Cacoub P, Gougis P. [Differences of characteristics and outcomes between cancer patients and patients with no active cancer hospitalised for a SARS-CoV-2 infection]. Bull Cancer. 2021 Jun;108(6):581-588. doi: 10.1016/j.bulcan.2021.03.004. Epub 2021 Mar 20. French. PMID 33966886